CLINICAL TRIAL: NCT01575015
Title: Intra-Operative Continuous Renal Replacement Therapy in Liver Transplantation: A Phase II Randomized Controlled Trial (INCEPTION)
Brief Title: Intraoperative Dialysis in Liver Transplantation
Acronym: INCEPTION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding.
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Sean M Bagshaw, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOFAPro00026047
Record Dates: First submitted 2012-03-25; First posted 2012-04-10 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Liver Failure; Acute Kidney Disease; Multi-organ Failure
Keywords: Liver transplantation (E04.210.650); Renal replacement therapy (E05.196.353); Intra-operative period (E04.614.374); Safety (N06.850.135.060.075); Efficacy
MeSH Terms: conditions — Liver Failure; Multiple Organ Failure | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard intraoperative support (no CRRT) (Active Comparator)
  Interventions: Procedure: Standard intraoperative support
- Intraoperative renal support (CRRT) (Experimental)
  Interventions: Device: Continuous renal replacement therapy (CRRT)

INTERVENTIONS:
Device: Continuous renal replacement therapy (CRRT) — Patients allocated with intraoperative CRRT will have a dialysis catheter inserted and receive CRRT during liver transplantation
  Arms: Intraoperative renal support (CRRT)
Procedure: Standard intraoperative support — Patients allocated to standard intraoperative support will receive usual care (no CRRT).
  Arms: Standard intraoperative support (no CRRT)

SUMMARY:
Patient with liver failure waiting for liver transplantation are often hospitalized and commonly supported in an intensive care unit prior to surgery. These patients are sick, and in addition to the complications of a failing liver, other organs such as the kidneys often fail as well. As a consequence, these patients are at an increased risk for complications related to their kidney failure during their liver transplantation procedure. One potential method to diminish the risk of these complications is to provide dialysis support to these patients during their liver transplantation in the operating theater in the form of continuous renal replacement therapy (CRRT). While this is increasingly being performed and is theoretically appealing, there is very little information to support this practice. In addition, the use of CRRT during surgery is not entirely without risk. The investigators have performed two preliminary studies on the use of CRRT during liver transplantation and our data would strongly support the need to conduct further higher-quality studies to better evaluate its feasibility, safety and usefulness. Our proposed study is for a randomized trial comparing the use of CRRT during surgery with standard supportive care in sick patients with liver failure scheduled to receive a liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* Adult (age > 18 years on the day of assessment of eligibility)
* Planned cadaveric orthotopic liver transplantation
* Pre-operative unadjusted (natural) Modification of End-Stage Liver Disease (MELD) score > 25.
* Pre-operative AKI, defined by a minimum RIFLE-RISK, AND/OR pre-operative estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, calculated by the Modification of Diet in Renal Disease (MDRD) equation.

Exclusion Criteria:

* Planned living-related donor liver transplantation
* Pre-operative potassium [K] > 4.5 mmol/L AND urine output < 100 mL in the 6 hrs preceding assessment of eligibility
* Pre-operative pH < 7.3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Number of patients adhering to the prescribed protocol | Intra-operative (From the induction of anesthesia to trasnfer from the OR to the ICU, average 6-8 hours)
  Will be defined as the proportion of patients adhering to the prescribed protocol.
Number of patients with adverse events | Intra-operative (From the induction of anesthesia to trasnfer from the OR to the ICU, average 6-8 hours)
  This will be defined by the proportion of patients experiencing intra-operative adverse events, serious adverse events and complications related to the study intervention.

SECONDARY OUTCOMES:
Fluid balance | In-hospital (patients will be followed for duration of post-operative hospital stay, anticipated average 4 weeks post-operatively)
  Will be defined as the changes in fluid accumulation intra- and post-operatively.
Number of patients with post-operative graft dysfunction | In-hospital (patients will be followed for duration of post-operative hospital stay, anticipated average 4 weeks post-operatively)
  Graft dysfunction will include post-operative ultrasonographic-evidence of vascular ischemia/occlusion or venous occlusion; biliary stricture, obstruction or anastomosis leak; primary non-function; biopsy-proven rejection; or need for surgical re-exploration for any reason.
Number of patients with post-operative kidney dysfunction | From the date of liver transplant until the date of first documented outcome of interest, assessed until 90-days
  Will be defined as post-operative acute kidney injury, defined by RIFLE criteria; along with encompassing receipt of renal replacement therapy (RRT).
Length of stay | From the date of liver transplant until the date of discharge from ICU/hospital
  Will include ICU and hospital lengths of stay
Mortality | From the date of liver transplant until the date of first documented outcome of interest, assessed until 90-days
  Mortality through 90-days.
Number of patients readmitted to hospital within 90-days | From the date of liver transplant after hospital discharge, until the date of first documented re-admission to hospital, assessed until 90-days
  Will be defined as hospital re-admission within 90-days of liver transplant for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Bagshaw, MD, MSc, Principal Investigator — Division of Critical Care Medicine, Faculty of Medicine and Dentistry, University of Alberta
Locations (1):
- Division of Critical Care Medicine, University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Townsend DR, Bagshaw SM, Jacka MJ, Bigam D, Cave D, Gibney RT. Intraoperative renal support during liver transplantation. Liver Transpl. 2009 Jan;15(1):73-8. doi: 10.1002/lt.21650. PMID 19109832
- [Background] Parmar A, Bigam D, Meeberg G, Cave D, Townsend DR, Gibney RT, Bagshaw SM. An evaluation of intraoperative renal support during liver transplantation: a matched cohort study. Blood Purif. 2011;32(3):238-48. doi: 10.1159/000329485. Epub 2011 Aug 9. PMID 21829016
- [Derived] Karvellas CJ, Taylor S, Bigam D, Kneteman NM, Shapiro AMJ, Romanovsky A, Gibney RTN, Townsend DR, Meeberg G, Ozelsel T, Bishop E, Bagshaw SM. Intraoperative continuous renal replacement therapy during liver transplantation: a pilot randomized-controlled trial (INCEPTION). Can J Anaesth. 2019 Oct;66(10):1151-1161. doi: 10.1007/s12630-019-01454-0. Epub 2019 Jul 26. PMID 31350701